CLINICAL TRIAL: NCT01799785
Title: Aerobic Training in Patients With Cirrhosis
Brief Title: Effects of Aerobic Training on Exercise Capacity in Patients With Cirrhosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Puneeta Tandon, Associate Professor Medicine, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LZPTMH1
Record Dates: First submitted 2013-02-08; First posted 2013-02-27 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerobic exercise (Experimental): Supervised aerobic training 3 times per week for 8 weeks (30-60 minute sessions)
  Interventions: Behavioral: Aerobic exercise
- Usual care group (Placebo Comparator): These patients will continue with their normal daily activity and will not be provided with supervised aerobic exercise training during the study period.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Aerobic exercise — Aerobic exercise for 8 weeks (3 times per week, 30-60 minutes each session)
  Arms: Aerobic exercise
Other: Usual Care
  Arms: Usual care group

SUMMARY:
Cirrhosis is associated with a reduction in muscle mass and exercise capacity. This has an impact or morbidity and mortality. Regular aerobic exercise training is a proven effective therapy to improve exercise capacity in healthy and clinical populations. the effect of this training has not yet been evaluated in cirrhosis. The safety of this intervention also requires further study. Using a randomized controlled design, the investigators aim to conduct a pilot study evaluating the safety and efficacy of eight weeks of aerobic exercise training on aerobic capacity.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤70 years
* Cirrhosis
* Child Pugh class A or B
* If required, primary or secondary variceal prophylaxis in place

Exclusion Criteria:

* Post-liver transplantation
* Hepatocellular carcinoma
* Active non-Hepatocellular carcinoma malignancy
* Significant cardiac disease - ejection fraction <60% or known coronary artery disease
* Oxygen saturation at rest <95%
* Known myopathy
* Hemoglobin (<100 g/L)
* Chronic renal failure on dialysis
* Physical impairment making it impossible to ride an exercise bike or treadmill
* Orthopedic abnormality preventing exercise training
* HIV infection
* Patient unwilling to consent to study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change in peak exercise pulmonary oxygen uptake (peak VO2) | Baseline (day 1) and Study End (8 weeks)

SECONDARY OUTCOMES:
Change in muscle mass as measured by thigh ultrasound | Baseline (day 1) and study end (8 weeks)
Change in Quality of Life - Chronic Liver Disease Questionnaire | Baseline (day 1) and Study End (8 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Haykowsky, Study Director — University of Alberta
Locations (1):
- University of Alberta, Mazankowski Heart Institute, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Zenith L, Meena N, Ramadi A, Yavari M, Harvey A, Carbonneau M, Ma M, Abraldes JG, Paterson I, Haykowsky MJ, Tandon P. Eight weeks of exercise training increases aerobic capacity and muscle mass and reduces fatigue in patients with cirrhosis. Clin Gastroenterol Hepatol. 2014 Nov;12(11):1920-6.e2. doi: 10.1016/j.cgh.2014.04.016. Epub 2014 Apr 24. PMID 24768811